CLINICAL TRIAL: NCT00000646
Title: Pentoxifylline (Trental) as a Modulator of Tumor Necrosis Factor and of HIV Replication in Patients With AIDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoechst Marion Roussel (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 160; 11135 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Pentoxifylline; Virus Replication; Tumor Necrosis Factor; Drug Evaluation; Acquired Immunodeficiency Syndrome; Cachexia; Drug Synergism
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Cachexia | interventions — Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline

SUMMARY:
To determine whether pentoxifylline lowers tumor necrosis factor (TNF) levels in AIDS patients. Pentoxifylline decreases tumor necrosis factor (TNF), and therefore should decrease such TNF-intensified events as cachexia, enhanced HIV expression, and inhibition of zidovudine (AZT) activity.

DETAILED DESCRIPTION:
Pentoxifylline decreases tumor necrosis factor (TNF), and therefore should decrease such TNF-intensified events as cachexia, enhanced HIV expression, and inhibition of zidovudine (AZT) activity.

Twenty-seven AIDS patients with elevated TNF and less than 300 CD4 cells are given pentoxifylline 3 times a day for 8 weeks. If no significant changes are seen in virologic, immunologic, or related measures, 27 additional patients are given a higher dose of pentoxifylline 3 times a day for eight weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Zidovudine (AZT), didanosine (ddI), dideoxycytidine (ddC), or a combination thereof, at current dosage for the 8 weeks of study treatment.
* Prophylaxis (e.g., aerosolized pentamidine, trimethoprim / sulfamethoxazole (TMP / SMX), dapsone for Pneumocystis carinii pneumonia (PCP) if CD4 cell count is < 200 cells/mm3

Allowed:

* Concurrent maintenance therapy for opportunistic infections.

Prior Medication: Required:

* Zidovudine (AZT), didanosine (ddI), dideoxycytidine (ddC), or a combination thereof, for at least 2 months.

Patients must have the following:

* Diagnosis of AIDS.
* Documented HIV seropositivity.
* Ability to give informed consent and willingness to comply with visit schedule and all procedures.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Lymphoma or visceral Kaposi's sarcoma.
* Active peptic ulcer or bleeding disorder.
* Hemophilia. Known intolerance to pentoxifylline, theophylline, or caffeine.

Concurrent Medication:

Excluded:

* Warfarin and heparin.
* Biological response modifiers (e.g., erythropoietin, interferon, G-CSF, GM-CSF).

Cytotoxic chemotherapy.

* Megestrol acetate. Corticosteroids.

Concurrent Treatment:

Excluded:

* Radiation therapy. Blood products or transfusions.

Patients with the following are excluded:

* Presence of an active opportunistic infection.
* Major surgery within 30 days of study treatment.

Prior Medication:

Excluded:

* Biological response modifiers (including interferon, interleukin), corticosteroids, or megestrol acetate within 14 days of first (screening) TNF level.
* Erythropoietin dependency or within 30 days of study treatment.

Prior Treatment:

Excluded:

* Transfusion or blood product dependency or use within 30 days of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Study Completion 1993-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dezube B, Study Chair; Crumpacker C, Study Chair
Locations (2):
- United States (2):
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Case CRS, Cleveland, Ohio

REFERENCES:
- [Background] Dezube BJ, Lederman MM, Pardee AB, Chapman B, Korvick J, Crumpacker CS. Pentoxifylline (Trental, PTX) decreases tumor necrosis factor (TNF) & may decrease HIV replication in AIDS patients. ACTG #160 Team. Int Conf AIDS. 1993 Jun 6-11;9(1):492 (abstract no PO-B28-2142)
- [Background] Dezube BJ, Pardee AB, Chapman B, Beckett LA, Korvick JA, Novick WJ, Chiurco J, Kasdan P, Ahlers CM, Ecto LT, et al. Pentoxifylline decreases tumor necrosis factor expression and serum triglycerides in people with AIDS. NIAID AIDS Clinical Trials Group. J Acquir Immune Defic Syndr (1988). 1993 Jul;6(7):787-94. PMID 8099612
- [Background] Dezube BJ, Pardee AB, Chapman B, Beckett L, Korvick J, Ahlers CM, Ecto L, Chatis P, Crumpacker CS. Pentoxifylline (trental) decreases tumor necrosis factor (TNF) and HIV replication in patients with AIDS. ACTG #160 Team. AIDS Clinical Trial Group. Int Conf AIDS. 1992 Jul 19-24;8(1):Mo8 (abstract no MoB 0019)
- [Background] Dezube BJ, Lederman MM, Spritzler JG, Chapman B, Korvick JA, Flexner C, Dando S, Mattiacci MR, Ahlers CM, Zhang L, et al. High-dose pentoxifylline in patients with AIDS: inhibition of tumor necrosis factor production. National Institute of Allergy and Infectious Diseases AIDS Clinical Trials Group. J Infect Dis. 1995 Jun;171(6):1628-32. doi: 10.1093/infdis/171.6.1628. PMID 7769305
- [Background] Dezube BJ, Pardee AB, Beckett LA, Ahlers CM, Ecto L, Allen-Ryan J, Anisowicz A, Sager R, Crumpacker CS. Cytokine dysregulation in AIDS: in vivo overexpression of mRNA of tumor necrosis factor-alpha and its correlation with that of the inflammatory cytokine GRO. J Acquir Immune Defic Syndr (1988). 1992;5(11):1099-104. PMID 1403638